CLINICAL TRIAL: NCT04222842
Title: Phase I Study of CM082 in Patients With Myopic Choroidal Neovascularization (CNV)
Brief Title: CM082 in Patients With Myopic Choroidal Neovascularization (CNV)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Day is not required for Anticipated dates.
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM082-OPH-I-102
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Myopic Choroidal Neovascularisation
MeSH Terms: interventions — vorolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM082 Tablet (Experimental): Code Name: CM082 Tablet Other Name: X-82 Dosage and Administration: 25mg BID/50mg QD/50mg BID, P.O., two-week on/two-week off in four-week cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CM082

INTERVENTIONS:
Drug: CM082 — Subjects will receive CM082 orally for two weeks followed by two weeks off in four-week cycles.The total treatment period is tentatively set at 3 cycles (12 weeks).
  Other Names: X-82

SUMMARY:
This is a Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Intermittent Oral Dosing of CM082 tablets in Chinese Patients With mCNV.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase I Study to Evaluate the safety, tolerability, pharmacokinetics and preliminary Efficacy of intermittent oral dosing of CM082 tablets in Chinese patients with mCNV. The study will be performed in two different parts, dose-escalation phase (Part 1) and dose-expansion phase (Part 2). Subjects will receive CM082 orally for two weeks followed by two weeks off in four-week cycles. There are three dose levels, 25mg BID,50mg QD and 50mg BID. The total treatment period is tentatively set at 3 cycles (12 weeks). Based on data from dose escalation studies, identify safe and effective doses for expanded enrollment studies.The assessment of the safety and efficacy will be done in 2、4、8、12weeks after the first dose.Also, single/multiple dose pharmacokinetics in these patients will be studied.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of active CNV secondary to pathologic myopia and the study eye must have the following lesion characteristics: (a)presence of high myopia with greater than -6 diopters of spherical equivalencef or anteroposterior elongation greater than 26 mm, (b) presence of at least 1 of the following lesion types: subfoveal; juxtafoveal; extrafoveal with involvement of the central macular area and margin of the optic disk with involvement of the central macular area, (c) vision loss due to the above causes, (d) ETDRS BCVA 24 to 78 letters.
* Patients with no previous anti-VEGF therapy.
* Adequate bone marrow, hepatic, and renal functions.
* Willing to sign the ICF and comply with the study protocol.

Exclusion Criteria:

* CNV due to causes other than mCNV.
* Any significant disease in the study eye that could compromise BCVA.
* Active eye infection in any eye.
* Previous treatment with photodynamic therapy (PDT), external beam radiation, laser photocoagulation, or transpupillary thermotherapy within

  1 month of the first dose.
* Intraocular surgery in the test eye within 3 months prior to the first dose.
* Any eye received intravitreal injection of corticosteroids within 3 months prior to first dose.
* Clinically significant, uncontrolled cardiovascular and cerebrovascular disease.
* Patients who had previously used strong inhibitors of CYP3A or strong inducers were discontinued from the first dose of CM082 <5 drug half-lives (except for withdrawals longer than 14 days).
* Active hepatitis B (serum HBV DNA ≥ 500 IU / ml), hepatitis C antibody positive, HIV antibody positive or syphilis antibody positive.
* Swallowing dysfunction, active gastrointestinal disease, or other diseases that affect the absorption, distribution, metabolism, and excretion of drugs.
* Use of any investigational agent or participation in any other clinical trial of an investigational agent or investigational therapy within thirty (30) days of the first dose.
* Allergy to the ingredients of the study drug.
* Patients who have fertility needs and who cannot use effective methods of contraception during the study period and at least 3 months after the end of treatment (except for male patients after birth control or female patients after birth control or postmenopausal).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity(DLT) | the first cycle(the first four weeks)
  Any serious adverse event in eye or any ≥3 grade adverse reactions cannot be reduced to below grade 3 after treatment for more than 7 days.
Adverse event | 12 weeks
  Incidence of the adverse event after treatment

SECONDARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) | 12 weeks
  Change from baseline in mean BCVA (ETDRS)
Change in Choroidal Neovascularization (CNV) size | 12 weeks
  Change from baseline in mean CNV size (FA)
Change in Central Retinal Thickness | 12 weeks
  Change from baseline in mean central retinal thickness (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China